CLINICAL TRIAL: NCT07343778
Title: A Single-Arm, Open-Label, Multicenter Phase III Clinical Trial to Evaluate the Safety of Hydronidone Capsules in Patients With Hepatic Fibrosis and Liver Cirrhosis
Brief Title: A Clinical Trial Evaluating the Safety of Hydronidone Capsules in Patients With Hepatic Fibrosis and Liver Cirrhosis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KDN-F351-202508
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Chronic Hepatitis B With Hepatic Fibrosis
Keywords: Chronic hepatitis B with hepatic fibrosis
MeSH Terms: interventions — hydronidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydronitone Capsules group (Experimental): Eligible subjects who passed screening were enrolled sequentially in this study and received Hydronidone Capsules 120mg TID for 28 consecutive days.
  Interventions: Drug: Hydronidone Capsules

INTERVENTIONS:
Drug: Hydronidone Capsules — 120mg TID for 28 consecutive days

SUMMARY:
This is a single-arm, multicenter, open-label Phase III clinical trial to evaluate the safety and tolerability of high-dose hydronidone capsules in patients with hepatic fibrosis and cirrhosis. Eligible participants will be sequentially enrolled to receive hydronidone capsules 120 mg three times daily (TID) for 28 consecutive days. Participants will return to the hospital on Day 28 after the first dose for a follow-up safety assessment. All adverse events (AEs) and concomitant medications must be recorded during the study period. Participants who complete the Day 28 follow-up visit are considered to have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants fully understand the study, voluntarily participate, and have signed the informed consent form (ICF).
* Aged ≥18 years, regardless of gender.
* Have a confirmed diagnosis of hepatic fibrosis or cirrhosis based on either:

A prior percutaneous liver biopsy (results within 1 year prior to enrollment are acceptable); or

Imaging findings (Fibroscan, Fibrotouch, or ultrasound, with results within 3 months prior to enrollment acceptable).

* Alanine aminotransferase (ALT) < 8 × upper limit of normal (ULN).
* Female participants of childbearing potential must have a negative serum pregnancy test. Furthermore, the participant or their partner must agree to employ highly effective contraceptive methods from the start of the trial until 6 months after the last dose of the study drug.

Exclusion Criteria:

* History of major upper gastrointestinal hemorrhage within the past 3 months prior to enrollment, or the presence of gastrointestinal disorders affecting drug absorption at the time of screening.
* Total bilirubin (TBIL) > 3 × upper limit of normal (ULN), or ALT > 3 × ULN but < 8 × ULN and TBIL > 2 × ULN.
* Alpha-Fetoprotein (AFP) > 100 μg/L, even in the absence of clinical indications of hepatocellular carcinoma.
* Platelet count (PLT) ≤ 50 × 10⁹/L; Prothrombin activity (PTA) < 50% or International Normalized Ratio (INR) > 1.5.
* Active bacterial, viral (excluding chronic viral hepatitis B or C), fungal, or parasitic infection within 4 weeks prior to screening, or any infectious event requiring systemic anti-infective therapy.
* Positive test for Human Immunodeficiency Virus antibody (HIV-Ab).
* History of definite malignant tumors, or clinically significant dysfunction of major organs including heart, lungs, or kidneys, as well as clinically significant severe hepatic dysfunction unrelated to the underlying liver disease (e.g., manifestations of decompensated cirrhosis).
* Pregnant or lactating women.
* Participation in any other clinical trial and receipt of investigational drugs within 3 months prior to screening.
* Any other condition deemed by the investigator as unsuitable for enrollment or likely to prevent completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Any adverse events occurring in study participants following drug administration. | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth People's Hospital of Zhengzhou City, Zhengzhou, China